CLINICAL TRIAL: NCT02149732
Title: An Investigator-initiated Trial (IIT) on the Effect of Autologous Oral Mucosal Epithelial Sheet Transplantation in Corneal Limbal Deficiency Patients
Brief Title: Clinical Trial on the Effect of Autologous Oral Mucosal Epithelial Sheet Transplantation
Status: Available | Type: Expanded Access
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor
Other Study IDs: COMET trial; MKKim (Other Grant/Funding Number: Ministry of Health & Welfare, Republic of Korea (HI11C1590))
Record Dates: First submitted 2014-05-14; First posted 2014-05-29 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Limbal Stem Cell Deficiency; Stevens-johnson Syndrome; Ocular Cicatricial Pemphigoid; Chemical Burn
Keywords: Limbal stem cell deficiency; Cultivated oral mucosal cell sheet transplantation; Ocular surface reconstruction
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Stevens-Johnson Syndrome; Pemphigoid, Benign Mucous Membrane; Burns, Chemical

INTERVENTIONS:
Biological: cultivated oral mucosal epithelial sheet transplantation — Autologous cultivated oral mucosal epithelial cell sheet transplantation using oral mucosal adult stem cells in the patients with intractable corneal limbal deficiency

SUMMARY:
To investigate the effect of ocular surface reconstruction and assess the safety in cultivated oral mucosal epithelial cell sheet transplantation (COMET) regarding patients with cicatricial change of ocular surface.

DETAILED DESCRIPTION:
Interventional study for treatment of patients with cicatricial change of ocular surface.

Single Group: (Limbal stem cell deficiency group)

Treatment: After cultivating autologous Oral mucosal epithelial cell sheet, the sheet will be transplanted to the ocular surface of the patients

Inclusion criteria

1. patient with eye which has limbal stem cell deficiency and conjunctivalization of cornea
2. patient who shows no improvement after limbal tissue or amniotic membrane transplantation, or who has difficulty in receiving long-term immunosuppressive treatment
3. patient who agree this clinical trial
4. patient with the eyes in which best corrected visual acuity is less than counting finger
5. patient who is older than sixteen year old

Exclusion criteria

1. patient who has relevant corneal transparency
2. patient who is on the pregnancy or has a plan of pregnancy within 1 year
3. patient who has corneal infection
4. patient who has diagnosis of HBV, HCV, HIV, syphilis
5. patinet who has past medial history of antinal, myocardial infarction, heart failure, arrhythmia, brain stroke, cerebrovascular disease
6. patient who has malignancy
7. patient who shows hypersensitivity to bovine protein.

Primary outcome Epithelization of corneal surface (6 months after cell sheet transplantation)

Secondary outcome Visual acuity (6 months after cell sheet transplantation)

ELIGIBILITY:
Inclusion Criteria:

1. patient with eye which has limbal stem cell deficiency and conjunctivalization of cornea
2. patient who shows no improvement after limbal tissue or amniotic membrane transplantation, or who has difficulty in receiving long-term immunosuppressive treatment
3. patient who agree this clinical trial
4. patient with the eyes in which best corrected visual acuity is less than counting finger
5. patient who is older than sixteen year old

Exclusion Criteria:

1. patient who has relevant corneal transparency
2. patient who is on the pregnancy or has a plan of pregnancy within 1 year
3. patient who has corneal infection
4. patient who has diagnosis of HBV, HCV, HIV, syphilis
5. patinet who has past medial history of antinal, myocardial infarction, heart failure, arrhythmia, brain stroke, cerebrovascular disease
6. patient who has malignancy
7. patient who shows hypersensitivity to bovine protein.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mee Kum Kim, MD, PhD, Principal Investigator — Department of Ophthalmology, Seoul National University College of Medicine
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, Seoul
  - Seoul National Unversity Hospital, Seoul, Seoul

REFERENCES:
- [Background] Nishida K, Yamato M, Hayashida Y, Watanabe K, Yamamoto K, Adachi E, Nagai S, Kikuchi A, Maeda N, Watanabe H, Okano T, Tano Y. Corneal reconstruction with tissue-engineered cell sheets composed of autologous oral mucosal epithelium. N Engl J Med. 2004 Sep 16;351(12):1187-96. doi: 10.1056/NEJMoa040455. PMID 15371576